CLINICAL TRIAL: NCT02286609
Title: A Single Dose Evaluation of the Effects of Moderate (Child-Pugh Grade B) Hepatic Impairment on Deflazacort Pharmacokinetics
Brief Title: A Single Dose Evaluation of the Effects of Moderate Hepatic Impairment on Deflazacort Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MP-104-CL-023
Record Dates: First submitted 2014-11-04; First posted 2014-11-10 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Hepatic Impairment
MeSH Terms: interventions — deflazacort

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hepatic Impairment (Experimental): Eight (8) subjects with moderate hepatic insufficiency (a score of 7 to 9, on the Child-Pugh scale) will receive one 18 mg dose of deflazacort
  Interventions: Drug: Deflazacort
- Healthy Volunteer (Experimental): Eight (8) healthy subjects. Subjects will be matched for age [± 15 years], BMI [± 15 %], and gender [1:1] to the subjects in the moderate hepatic impaired cohort; will receive 18 mg dose of deflazacort
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Deflazacort — Deflazacort, a glucocorticoid with anti-inflammatory and immunosuppressive effects, is used in treating a variety of diseases. Pharmacologically it is an inactive pro-drug which is metabolized immediately to the active metabolite, 21 desacetyl-DFZ. The elimination of this metabolite is primarily via the urine in humans. Its potency is approximately 70 to 90% of prednisone and 6 mg of deflazacort has approximately the same anti-inflammatory potency as 5 mg of prednisolone or prednisone.
  Other Names: DFZ

SUMMARY:
This is a non-randomized, open-label, single-dose study to compare the PK of 21-desacetyl-DFZ and, if data permits, deflazacort in 8 subjects with moderate hepatic impairment (based on the Child Pugh classification, Grade B) to that of 8 healthy matched control subjects (age, body mass index [BMI], and gender).

DETAILED DESCRIPTION:
This is a non-randomized, open-label, single-dose study to compare the PK of 21-desacetyl-DFZ and, if data permits, deflazacort in 8 subjects with moderate hepatic impairment (based on the Child Pugh classification, Grade B) to that of 8 healthy matched control subjects (age, body mass index [BMI], and gender).

On Day 1, a single oral dose of deflazacort will be administered followed by serial blood sampling for 24 hours to assess the PK of 21-desacetyl-DFZ and, if data permits, deflazacort.

Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

Subjects will return to the Clinical Research Unit (CRU) 3 days (± 1 day) following study drug administration to determine if any adverse events (AEs) have occurred since the last study visit. Subjects who terminate the study early will be contacted if the Principal Investigator (PI) deems necessary.

A total of sixteen (16) adult male and female subjects will be enrolled. Hepatic Impaired Cohort: Eight (8) subjects with moderate hepatic insufficiency (a score of 7 to 9, on the Child-Pugh scale).

Healthy Match Control Cohort: Eight (8) healthy subjects. Subjects will be matched for age [± 15 years], BMI [± 15 %], and gender [1:1] to the subjects in the moderate hepatic impaired cohort.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Continuous non-smokers or moderate smokers.
* For a female of non-childbearing potential: must have undergone one a sterilization procedures or be postmenopausal with amenorrhea for at least 1 year prior to dosing and FSH serum levels consistent with postmenopausal status
* A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days
* If male, must agree not to donate sperm from dosing until 90 days Subject with Moderate Hepatic Impairment
* Adult male or female, 18 80 years of age
* BMI ≥ 18.5 and ≤ 40.0 kg/m2
* Subject's score on the Child-Pugh scale must range from 7 to 9 (moderate hepatic insufficiency)
* Subject has a diagnosis of chronic (> 6 months), stable (no acute episodes of illness within the previous 2 months due to deterioration in hepatic function) hepatic insufficiency with features of cirrhosis due to any etiology.

Healthy Subject

- Healthy adult male and female subjects will be matched 1:1 to a specific subject in the moderate hepatic impairment cohort based upon age, BMI, and gender.

Exclusion Criteria:

* Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug, related compounds (e.g., steroids or their formulations including lactose and corn starch).
* History (within the last year prior to dosing) or presence of peptic ulcers.
* History or presence of:

  * Gastritis or esophagitis, diverticulitis, ulcerative colitis (if there is probability of impending perforation), abscess or pyogenic infections, or fresh intestinal anastomosis;
  * Previous corticoids-induced myopathy;
  * Ocular herpes simplex;
  * Symptomatic cardiomyopathy at screening;
  * Immunosuppression or other contraindications for corticosteroid treatment;
  * History of chronic systemic fungal or viral infections;
  * Galactose intolerance, Lapp lactose deficiency, or glucose-galactose malabsorption;
  * Osteoporosis;
  * Myasthenia gravis;
  * Epilepsy;
  * Idiopathic hypocalcuria.
* Seated blood pressure is less than 90/40 mmHg or greater than 160/95 mmHg
* Seated heart rate is lower than 40 bpm or higher than 99 bpm
* QTcF interval is > 500 msec
* Has received any live or live-attenuated vaccine within 30 days
* Has received any immunosuppressive agents, coal tar, and/or radiation therapies within 30 days
* Has received injectable corticoids in the 12 weeks prior to dosing or any oral form of corticoids in 30 days
* Unable to refrain from or anticipates the use of:

  * Any drug known to be moderate or strong inhibitors or inducers of cytochrome P450 (CYP) 3A or P-glycoprotein (P-gp) for 14 days or 28 days, respectively
  * Any medication or substance, vitamin supplements, natural or herbal supplements which cannot be discontinued at least 14 days
* Female subjects of childbearing potential.
* Female subjects who are pregnant or lactating.
* Positive results at screening for HIV.
* Has been on a diet incompatible with the on study diet within 28 days
* Donation of blood or significant blood loss within 56 days
* Plasma donation within 7 days
* Participation in another clinical trial within 28 days Subject with Moderate Hepatic Impairment
* Has history of organ transplant.
* History of drug abuse within the past 2 years
* Has a positive urine drug or urine/breath alcohol testing Healthy Subject
* History or presence of alcoholism or drug abuse within the past 2 years
* Positive urine drug or urine/breath alcohol testing results at screening or check in.
* Positive results at screening for HBsAg or HCV.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Hepatic impairment on the pharmacokinetics (PK) of deflazacort in subjects with moderate hepatic impairment including the area under the plasma concentration time curve, from time 0 to the last measurable non-zero concentration. | 1 day
  Hepatic impairment on the pharmacokinetics (PK) of deflazacort in subjects with moderate hepatic impairment including the area under the plasma concentration time curve, from time 0 to the last measurable non-zero concentration.

SECONDARY OUTCOMES:
Safety and tolerability of one dose of deflazacort in subjects with hepatic impairment as measured by capturing occurrence of adverse events. | 1 day
  Safety and tolerability of one dose of deflazacort in subjects with hepatic impairment as measured by capturing occurrence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Bioscience Center, Study Director — Marathon Pharmaceuticals, LLC
Locations (2):
- United States (2):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida